CLINICAL TRIAL: NCT07082621
Title: Effectiveness of N Acetylcystene in Treatment of Radiotherapy Induced Oral Mucositis in Oral Cancer Patients (A Randomized Controlled Clinical Trial)
Brief Title: N Acetylcystene in Treatment of Radiotherapy Induced Oral Mucositis in Oral Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0727072023
Record Dates: First submitted 2025-07-12; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental)
  Interventions: Drug: N-acetylcysteine (NAC) spray
- Control Group (Active Comparator)
  Interventions: Drug: Conventional treatment

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) spray — N-acetylcysteine (NAC) mucoadhesive nanoparticles in the form of spray 3 times daily for 6 weeks
  Arms: Test Group
Drug: Conventional treatment — topical anesthetics agents (BBC [Benzocaine, Benzydamine, and Cetalkonium chloride] oral spray - oracure gel), topical antifungal agents (Miconaz oral gel)*, sodium bicarbonate mouth wash (Alkamsir sachets), ice chip,s and anti-inflammatory mouth wash.
  (Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology [MASCC/ISSO] guidelines) 3 times daily for 6 weeks.
  Arms: Control Group

SUMMARY:
Background: Radiotherapy appears to be one of the most effective therapies in head and neck tumors, however, there are a lot of complications related to it. Oral Mucositis is one of the most common complications following radiotherapy. There are currently huge unmet needs for management of oral mucositis. It causes severe pain, reduces food intake and affects quality of life of the head and neck cancer patients .N-acetylcysteine (NAC) is a glutathione precursor which has an antioxidant property and protects against radiation therapy-induced free radical damage. NAC reduces the production of inflammatory markers which leads to decrease inflammation, treats oral mucositis and enhances quality of life of the patient. Aim: To evaluate the effectiveness of N-acetylcysteine and its formulated nanoparticles in treatment of radiotherapy induced oral mucositis in oral cancer patients .

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with oral cancer by incisional biopsy histological examination.
* Patients above the age of 20 years.
* Patients receiving radiotherapy either as postoperatory (adjuvant) or as a definitive therapy in the treatment for oral cancer.
* Patients with radiotherapy induced-oral mucositis.
* Radiation dose ≥ 60 Gy which is responsible for oral mucositis development in oral cancer patients.

Exclusion Criteria:

* Patients diagnosed with any other type of cancer.
* Patients with any systemic disease as diabetes, cardiovascular, liver disorders and kidney disorders.
* Patients under anticoagulants such as warfarin, heparin or aspirin.
* Patients with findings of any physical or mental abnormalities

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-09 (Actual)

PRIMARY OUTCOMES:
Change in pain scores | Baseline,1,2,4,6 weeks
  The Numerical Rating Scale (NRS-11):- where patients are asked to rate their pain on a scale of 0 to 10 where 0 is no pain and 10 is the worst possible pain
change in oral mucositis severity | Baseline and 6 weeks
  Oral mucositis assessment scale (OMAS ) will be used to detect severity of oral mucositis at different mucosal sites in cm2 For each site, erythema is graded from 0 to 2 (none to severe), and ulceration/pseudomembrane formation is graded from 0 to 3 (none to >3 cm²).

SECONDARY OUTCOMES:
Serum gastrin 17 | Baseline and 6 weeks
  It will be measured at baseline and after 6 weeks by collecting fasting blood samples and analyzed by enzyme immunoassay 201-12-2036 human Gastrin(GAS) ELISA kit (96T) as directed by the manufacturer
Change in patient quality of life | Baseline and 6 weeks
  Oral health impact profile 14 (OHIP-14):- 14 questions, 0-4 score per question, range 0-14) questionnaires will be used to assess the effect of N -acetyl cysteine application on any change in subjective symptoms and quality of life as experienced by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral medicine Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt